CLINICAL TRIAL: NCT03397706
Title: A Phase 1b/2 Open-Label, Dose Escalation & Expansion Study of Orally Administered Viracta (VRx)-3996 & Valganciclovir in Subjects With Epstein-Barr Virus-Associated Lymphoid Malignancies
Brief Title: Dose Escalation & Expansion Study of Oral VRx-3996 & Valganciclovir in Subjects With EBV+ Lymphoid Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Viracta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VT3996-201
Record Dates: First submitted 2017-12-20; First posted 2018-01-12 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Epstein-Barr Virus-Associated Lymphoma; Lymphoproliferative Disorders
Keywords: EBV-associated peripheral T-cell lymphoma; EBV-associated angioimmunoblastic T-cell lymphoma; EBV-associated diffuse large B-cell lymphoma; EBV-associated post-transplant lymphoproliferative disorder; EBV-associated extranodal NK/T-cell lymphoma; EBV-associated Hodgkin lymphoma; EBV-associated non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoproliferative Disorders | interventions — Valganciclovir; Ganciclovir; 2-(6-(((6-fluoroquinolin-2-yl)methyl)amino)bicyclo(3.1.0)hex-3-yl)-N-hydroxypyrimidine-5-carboxamide

STUDY DESIGN:
Intervention Model Description: Phase 1: dose escalation phase (3+3 design with definitions of dose limiting toxicity) to define a recommended phase 2 dose
  Phase 2: dose expansion
  Tablet PK Cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1b Dose Escalation (Experimental): VRx-3996 (cohort 1) and valganciclovir
  VRx-3996 (cohort 2) and valganciclovir
  VRx-3996 (cohort 3) and valganciclovir
  VRx-3996 (cohort 4) and valganciclovir
  VRx-3996 (cohort 5) and valganciclovir
  Interventions: Combination Product: VRx-3996 and valganciclovir
- Phase 2 Expansion - Capsule (Experimental): VRx-3996 and valganciclovir at the recommended Phase 2 dose (RP2D)
  Interventions: Combination Product: VRx-3996 and valganciclovir
- Phase 2 Expansion - Tablet (Experimental): VRx-3996 and valganciclovir at the recommended Phase 2 dose (RP2D)
  Interventions: Combination Product: VRx-3996 and valganciclovir

INTERVENTIONS:
Combination Product: VRx-3996 and valganciclovir — second-generation histone deacetylase (HDAC) inhibitor, nanatinostat (previously referred to as either VRx-3996 or CHR-3396)
  Other Names: nanatinostat; ganciclovir; Chroma (CHR)-3996

SUMMARY:
A two part, Phase 1b/2 study to define a recommended Phase 2 dose of VRx-3996 in combination with valganciclovir (Phase 1b) designed to evaluate the efficacy of this combination in relapsed/refractory Epstein-Barr Virus Associated Lymphoma (EBV+ lymphomas).

DETAILED DESCRIPTION:
The purpose of this study is to determine whether VRx-3996 in combination with valganciclovir is safe, determine the side effect profile, and to determine whether this therapy may help patients with EBV-related lymphomas. The study has two phases. Goals of the first phase include determining a safe and tolerable dose that can be administered in phase 2. Goals of the second phase include further evaluating the safety and tolerability of VRx-3996 in combination with valganciclovir, evaluating how the drugs are metabolized in the body, evaluating response rates and other exploratory objectives that will help the researchers evaluate how these drugs work in the body. Participants will receive daily oral doses of the two study drugs and will have multiple study visits where they will have blood collected, physical examinations, and other medical monitoring. Following completion of the Ph2, the study will enroll additional patients into a Tablet Pharmacokinetic (PK) cohort to investigate the PK parameters of the tablet formulation.

ELIGIBILITY:
Key Inclusion Criteria:

* Relapsed/refractory, pathologically confirmed Epstein-Barr Virus positive (EBV+) lymphoid malignancy or lymphoproliferative disease
* Absence of available therapy with reasonable likelihood of cure or significant clinical benefit
* Adequate hematologic, hepatic and renal function as defined by laboratory assessment

Key Exclusion Criteria:

* Known primary central nervous system (CNS) lymphoma
* Known CNS metastases or leptomeningeal disease unless appropriately treated and neurologically stable for at least 4 weeks
* Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
* Refractory graft versus host disease (GvHD) not responding to treatment
* Known active hepatitis B virus infection
* Circulating hepatitis C virus on quantitative polymerase chain reaction (qPCR)
* Known history of human herpes virus (HHV)-6 chromosomal integration
* Known history of HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill DeFratis Robinson, Study Director — Viracta Therapeutics
Locations (28):
- United States (22):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - UC Irvine Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Anschutz Cancer Pavilion, Aurora, Colorado
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - ASCLEPES Research Centers, Weeki Wachee, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Ruth M Rothstein CORE Center, Chicago, Illinois
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - The University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - St. Vincent Healthcare Cancer Center, Billings, Montana
  - John Theurer Cancer Center at Hackensack UMC, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - The Ohio State University Wexner Medical Center James Cancer Hospital, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Texas Oncology - Baylor Sammons Cancer Center, Dallas, Texas
- Brazil (6):
  - Centro de Hematologia e Oncologia da Bahia (CEHON), Salvador, Estado de Bahia
  - Hospital de Cancer de Pernambuco (HCP), Recife, Pernambuco
  - Hospital do Cancer Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Real e Benemerita Associacao Portuguesa de Beneficencia, São Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (HC-FMUSP), São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haverkos B, Alpdogan O, Baiocchi R, Brammer JE, Feldman TA, Capra M, Brem EA, Nair S, Scheinberg P, Pereira J, Shune L, Joffe E, Young P, Spruill S, Katkov A, McRae R, Royston I, Faller DV, Rojkjaer L, Porcu P. Targeted therapy with nanatinostat and valganciclovir in recurrent EBV-positive lymphoid malignancies: a phase 1b/2 study. Blood Adv. 2023 Oct 24;7(20):6339-6350. doi: 10.1182/bloodadvances.2023010330. PMID 37530631
- See also: Viracta Therapeutics, Inc. — http://www.viracta.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Starting valganciclovir dosage reductions based on creatinine clearance were allowed for participants with renal impairment.
Groups:
- Phase 1b Dose Escalation Cohort 1: Viracta (VRx)-3996: 10 mg twice daily (BID) valganciclovir: 900 mg BID
- Phase 1b Dose Escalation Cohort 2a: VRx-3996: 5 mg BID valganciclovir: 450 mg BID
- Phase 1b Dose Escalation Cohort 2b: VRx-3996: 10 mg once daily (QD) valganciclovir: 450 mg BID
- Phase 1b Dose Escalation Cohort 2c: VRx-3996: 10 mg QD valganciclovir: 900 mg QD
- Phase 1b Dose Escalation Cohort 3: VRx-3996: 20 mg QD on Days 1 to 4/week valganciclovir: 900 mg QD
- Phase 2 Dose Expansion - Capsule: VRx-3996 recommended Phase 2 dose [RP2D]: 20 mg once daily [QD] on Days 1 to 4/week) and valganciclovir 900 mg QD
- Phase 2 Expansion - Tablet: VRx-3996 recommended Phase 2 dose [RP2D]: 20 mg once daily [QD] on Days 1 to 4/week and valganciclovir 900 mg QD
Period: Overall Study
Arm/Group | Phase 1b Dose Escalation Cohort 1 | Phase 1b Dose Escalation Cohort 2a | Phase 1b Dose Escalation Cohort 2b | Phase 1b Dose Escalation Cohort 2c | Phase 1b Dose Escalation Cohort 3 | Phase 2 Dose Expansion - Capsule | Phase 2 Expansion - Tablet
Started | 7 | 5 | 4 | 4 | 5 | 30 | 9
Completed | 7 | 5 | 4 | 4 | 5 | 30 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Starting valganciclovir dosage reductions based on creatinine clearance were allowed for participants with renal impairment.
Groups:
- Phase 1b Dose Escalation Cohort 1: VRx-3996: 10 mg twice daily (BID) valganciclovir: 900 mg BID
- Phase 2 Dose Expansion - Capsule; Phase 2 Dose Expansion - Tablet: VRx-3996 (RP2D: 20 mg QD on Days 1 to 4/week) and valganciclovir (RP2D: 900 mg QD)
- Total: Total of all reporting groups
Arm/Group | Phase 1b Dose Escalation Cohort 1 | Phase 1b Dose Escalation Cohort 2a | Phase 1b Dose Escalation Cohort 2b | Phase 1b Dose Escalation Cohort 2c | Phase 1b Dose Escalation Cohort 3 | Phase 2 Dose Expansion - Capsule | Phase 2 Dose Expansion - Tablet | Total
Number analyzed (Participants) | 7 | 5 | 4 | 4 | 5 | 30 | 9 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 4 | 3 | 4 | 14 | 3 | 34
  >=65 years | 3 | 3 | 0 | 1 | 1 | 16 | 6 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (24.06) | 60.8 (20.44) | 45.3 (19.45) | 56.8 (10.56) | 44.0 (24.36) | 60.1 (16.97) | 63.4 (15.42) | 57.7 (18.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 1 | 2 | 12 | 4 | 24
  Male | 6 | 3 | 2 | 3 | 3 | 18 | 5 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 2 | 8 | 1 | 12
  Not Hispanic or Latino | 7 | 5 | 4 | 3 | 3 | 22 | 7 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 5
  White | 6 | 4 | 2 | 3 | 3 | 24 | 8 | 50
  More than one race | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 5 | 4 | 3 | 3 | 20 | 9 | 51
  Brazil | 0 | 0 | 0 | 1 | 2 | 10 | 0 | 13
Lymphoma or Lymphoproliferative Disorder Subtype [Count of Participants; unit: Participants]
  Peripheral T-cell Lymphoma / Angioimmunoblastic T-cell Lymphoma | 1 | 2 | 1 | 0 | 0 | 7 | 2 | 13
  Diffuse Large B-cell Lymphoma | 1 | 1 | 0 | 0 | 0 | 5 | 3 | 10
  Extranodal NK/T-cell Lymphoma | 0 | 0 | 1 | 0 | 2 | 6 | 1 | 10
  Human Immunodeficiency Virus-Associated Lymphoma | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 5
  Hodgkin Lymphoma | 2 | 0 | 0 | 1 | 1 | 7 | 1 | 12
  Immunodeficiency-Associated Lymphoproliferative Disorders | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 4
  Other B-cell Non-Hodgkin Lymphomas | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 4
  Other T-cell Non-Hodgkin Lymphomas | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Post-Transplant Lymphoproliferative Disorders | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number (Proportion) of Participants With Adverse Events (AEs)
Description: Number (percentage) of patients experiencing at least one treatment-emergent adverse event, defined as those untoward medical events with onset after the first dose of study drug or existing events that worsened after the first dose during the study
Time Frame: Up to approximately 2 years
Population: Safety Analysis Set, defined as all enrolled patients who received at least 1 dose of study treatment. Valganciclovir dosage reductions were allowed for participants with renal impairment at study entry or during study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Dose Escalation Cohort 1 | Phase 1b Dose Escalation Cohort 2a | Phase 1b Dose Escalation Cohort 2b | Phase 1b Dose Escalation Cohort 2c | Phase 1b Dose Escalation Cohort 3 | Phase 2 Dose Expansion - Capsule | Phase 2 Dose Expansion - Tablet
Number analyzed (Participants) | 7 | 5 | 4 | 4 | 5 | 30 | 9
Participants | 7 | 5 | 4 | 4 | 5 | 30 | 9

2. Primary Outcome: Number (Proportion) of Participants With Dose-Limiting Toxicities (DLTs) in Phase 1b
Description: Number (percentage) of patients experiencing a DLT during the first cycle (28 days) of study treatment in Phase 1b, defined as an adverse event (AE) or clinically significant abnormal laboratory value that was at least possibly related to study drugs and was not primarily related to disease, disease progression, concomitant medication(s), or intercurrent illness. In addition, to be considered a DLT, the AE had to meet at least one of the following criteria:
  * Grade 4 anemia unexplained by underlying disease
  * Grade 4 febrile neutropenia
  * Grade 4 neutropenia lasting >5 days
  * Any other Grade 4 hematologic toxicity (thrombocytopenia, neutropenia, febrile neutropenia, anemia) of any duration
  * Grade 4 or higher tumor lysis syndrome
  * Grade 3 or higher thrombocytopenia (with or without bleeding)
  * Any requirement for platelet transfusion
  * Grade 3 or higher non-hematologic toxicity despite adequate supportive care
  * Results in a dose hold of >7 consecutive days
Time Frame: Cycle 1 (28 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b Dose Escalation Cohort 3 (RP2D): VRx-3996: 20 mg QD on Days 1 to 4/week valganciclovir: 900 mg QD
Arm/Group | Phase 1b Dose Escalation Cohort 1 | Phase 1b Dose Escalation Cohort 2a | Phase 1b Dose Escalation Cohort 2b | Phase 1b Dose Escalation Cohort 2c | Phase 1b Dose Escalation Cohort 3 (RP2D)
Number analyzed (Participants) | 7 | 5 | 4 | 4 | 5
Participants | 4 | 0 | 0 | 0 | 0

3. Primary Outcome: Overall Response Rate
Description: Number (percentage) of patients with a best overall complete response (CR) or partial response (PR) according to the Lugano 2014 criteria (Cheson, Bruce D. et al. J Clin Oncology 2014;32(27):3059-68), where CR included complete metabolic response (no/minimal fluorodeoxyglucose [FDG] uptake) and radiologic response (target lesions regress to ≤1.5 cm in longest transverse diameter of a lesion) and no new lesions, and PR included partial metabolic response (reduced FDG uptake compared with baseline) or radiologic response (target lesions ≤ 50% decrease in the sum of the product of perpendicular diameters of up to 6 target measurable nodes and extranodal sites)
Time Frame: Up to approximately 2 years
Population: Efficacy Evaluable Analysis Set, defined as all patients with measurable/evaluable disease at screening who met all eligibility criteria and had at least one evaluable post-baseline efficacy tumor assessment. Valganciclovir dosage reductions were allowed for participants with renal impairment at study entry or during study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Dose Escalation Cohort 1 | Phase 1b Dose Escalation Cohort 2a | Phase 1b Dose Escalation Cohort 2b | Phase 1b Dose Escalation Cohort 2c | Phase 1b Dose Escalation Cohort 3 | Phase 2 Dose Expansion - Capsule | Phase 2 Dose Expansion - Tablet
Number analyzed (Participants) | 6 | 2 | 2 | 4 | 5 | 23 | 8
Participants
  Complete Response | 2 | 1 | 0 | 0 | 1 | 3 | 1
  Partial Response | 1 | 1 | 1 | 0 | 2 | 4 | 1
  Stable Disease | 1 | 0 | 0 | 1 | 1 | 5 | 1
  Progressive Disease | 2 | 0 | 1 | 3 | 1 | 11 | 5

4. Secondary Outcome: Duration of Response
Description: Interval of time from date of first observed complete or partial response per Lugano 2014 criteria (Cheson BD et al. J Clin Oncology 2014;32(27):3059-68) to the date of documented disease progression or death due to any cause, where disease progression is defined by Lugano 2014 criteria (Cheson BD et al. J Clin Oncology 2014;32(27):3059-68) as progressive metabolic disease (increase in fluorodeoxyglucose [FDG] uptake from baseline or new FDG-avid foci consistent with lymphoma) or progressive radiologic response (increase in the product of perpendicular diameters of a single node by ≥ 50% or emergence of a new lesion)
Time Frame: Up to approximately 2 years
Population: Patients who achieved a CR or PR. Valganciclovir dosage reductions were allowed for participants with renal impairment at study entry or during study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1b Dose Escalation Cohort 1 | Phase 1b Dose Escalation Cohort 2a | Phase 1b Dose Escalation Cohort 2b | Phase 1b Dose Escalation Cohort 2c | Phase 1b Dose Escalation Cohort 3 | Phase 2 Dose Expansion - Capsule | Phase 2 Dose Expansion - Tablet
Number analyzed (Participants) | 3 | 2 | 1 | 0 | 3 | 7 | 2
days | 825.5 [160.0 to NA] — The upper bound of the 95% confidence interval was not reached due to insufficient number of participants with events. | 116.5 [34.0 to NA] — The upper bound of the 95% confidence interval was not reached due to insufficient number of participants with events. | 113.0 [NA to NA] — The lower and upper bounds of the 95% confidence interval were not reached due to insufficient number of participants with events. |  | NA [127.0 to NA] — The median and upper bound of the 95% confidence interval were not reached due to insufficient number of participants with events. | 634.0 [80.0 to NA] — The upper bound of the 95% confidence interval was not reached due to insufficient number of participants with events. | NA [57.0 to NA] — The median and upper bound of the 95% confidence interval were not reached due to insufficient number of participants with events.

5. Secondary Outcome: Time to Response
Description: Interval of time from the start of study drug treatment to the first documentation of CR or PR per Lugano 2014 criteria (Cheson BD et al. J Clin Oncology 2014;32(27):3059-68)
Time Frame: Up to approximately 2 years
Population: Patients who achieved a PR or CR. Valganciclovir dosage reductions were allowed for participants with renal impairment at study entry or during study treatment.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Phase 2 Expansion - Capsule; Phase 2 Expansion - Tablet: VRx-3996 (RP2D: 20 mg QD on Days 1 to 4/week) and valganciclovir (RP2D: 900 mg QD)
Arm/Group | Phase 1b Dose Escalation Cohort 1 | Phase 1b Dose Escalation Cohort 2a | Phase 1b Dose Escalation Cohort 2b | Phase 1b Dose Escalation Cohort 2c | Phase 1b Dose Escalation Cohort 3 | Phase 2 Expansion - Capsule | Phase 2 Expansion - Tablet
Number analyzed (Participants) | 3 | 2 | 1 | 0 | 3 | 7 | 2
days | NA [33.0 to NA] — The median and upper bound of the 95% confidence interval were not reached due to insufficient number of participants with events. | 52.5 [51.0 to NA] — The upper bound of the 95% confidence interval was not reached due to insufficient number of participants with events. | NA [50.0 to NA] — The median and upper bound of the 95% confidence interval were not reached due to insufficient number of participants with events. |  | NA [57.0 to NA] — The median and upper bound of the 95% confidence interval were not reached due to insufficient number of participants with events. | 162.0 [58.0 to NA] — The upper bound of the 95% confidence interval was not reached due to insufficient number of participants with events. | NA [58.0 to NA] — The median and upper bound of the 95% confidence interval were not reached due to insufficient number of participants with events.

6. Secondary Outcome: Progression-Free Survival
Description: Interval of time from the date of first study drug administration to the documented date of disease progression or death, whichever occurred first, where disease progression is defined by Lugano 2014 criteria (Cheson BD et al. J Clin Oncology 2014;32(27):3059-68) as progressive metabolic disease (increase in fluorodeoxyglucose [FDG] uptake from baseline or new FDG-avid foci consistent with lymphoma) or progressive radiologic response (increase in the product of perpendicular diameters of a single node by ≥ 50% or emergence of a new lesion)
Time Frame: Up to approximately 2 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1b Dose Escalation Cohort 1 | Phase 1b Dose Escalation Cohort 2a | Phase 1b Dose Escalation Cohort 2b | Phase 1b Dose Escalation Cohort 2c | Phase 1b Dose Escalation Cohort 3 | Phase 2 Expansion - Capsule | Phase 2 Expansion - Tablet
Number analyzed (Participants) | 6 | 2 | 2 | 4 | 5 | 23 | 8
days | 209.0 [57.0 to NA] — The upper bound of the 95% confidence interval was not reached due to insufficient number of participants with events. | 168.0 [87.0 to NA] — The upper bound of the 95% confidence interval was not reached due to insufficient number of participants with events. | 107.5 [53.0 to NA] — The upper bound of the 95% confidence interval was not reached due to insufficient number of participants with events. | 55.5 [15.0 to NA] — The upper bound of the 95% confidence interval was not reached due to insufficient number of participants with events. | 185.0 [10.0 to NA] — The upper bound of the 95% confidence interval was not reached due to insufficient number of participants with events. | 66.0 [56.0 to 220.0] | 52.5 [34.0 to 114.0]

7. Secondary Outcome: Disease Control Rate
Description: Number (percentage) of patients with CR, PR, or stable disease (SD) per Lugano 2014 criteria (Cheson BD et al. J Clin Oncology 2014;32(27):3059-68)
Time Frame: Up to approximately 2 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Dose Escalation Cohort 1 | Phase 1b Dose Escalation Cohort 2a | Phase 1b Dose Escalation Cohort 2b | Phase 1b Dose Escalation Cohort 2c | Phase 1b Dose Escalation Cohort 3 | Phase 2 Expansion - Capsule | Phase 2 Expansion - Tablet
Number analyzed (Participants) | 6 | 2 | 2 | 4 | 5 | 23 | 8
Participants | 4 | 2 | 1 | 1 | 4 | 12 | 3

8. Secondary Outcome: Overall Survival
Description: Interval of time from date of first study drug treatment to date of death, for any reason (patients without documentation of death at the time of analysis were censored at the date the patient was last known to be alive)
Time Frame: Up to approximately 2 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1b Dose Escalation Cohort 1 | Phase 1b Dose Escalation Cohort 2a | Phase 1b Dose Escalation Cohort 2b | Phase 1b Dose Escalation Cohort 2c | Phase 1b Dose Escalation Cohort 3 | Phase 2 Expansion - Capsule | Phase 2 Expansion - Tablet
Number analyzed (Participants) | 6 | 2 | 2 | 4 | 5 | 23 | 8
days | 227.0 [122.0 to NA] — The upper bound of the 95% confidence interval was not reached due to insufficient number of participants with events. | 578.0 [486.0 to NA] — The upper bound of the 95% confidence interval was not reached due to insufficient number of participants with events. | NA [328.0 to NA] — The median and upper bound of the 95% confidence interval were not reached due to insufficient number of participants with events. | 168.5 [32.0 to NA] — The upper bound of the 95% confidence interval was not reached due to insufficient number of participants with events. | 496.0 [49.0 to NA] — The upper bound of the 95% confidence interval was not reached due to insufficient number of participants with events. | 801.0 [315.0 to NA] — The upper bound of the 95% confidence interval was not reached due to insufficient number of participants with events. | NA [106.0 to NA] — The median and upper bound of the 95% confidence interval were not reached due to insufficient number of participants with events.

9. Secondary Outcome: Cmax (ng/mL) of VRx-3996
Description: Pharmacokinetic (PK) assessment of VRx-3996 pre-dose and at hours 0.5, 1, 2, 4, and 6 post-dose on cycle 1 day 1 (C1D1) and cycle 2 day 2 (C2D1)
Time Frame: Phase 1b: Cycle 1 Day 1 and Phase 2: multiple doses through Cycle 2 Day 1
Population: The PK Analysis Set was used for all PK analyses and included all patients in the intent-to-treat population (defined as all enrolled patients) who had at least one postdose measurable PK concentration. The PK Analysis Set will be used for individual plasma concentration listings and summaries of plasma concentrations.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Phase 1b Dose Escalation Cohorts 1, 2b and 2c: VRx-3996: 10 mg QD or BID valganciclovir: 450 mg QD or BID or 900 mg QD or BID
- Phase 2 RP2D - Capsule; Phase 2 RP2D - Tablet: VRx-3996: 20 mg QD on Days 1 to 4/week valganciclovir: 900 mg QD
Arm/Group | Phase 1b Dose Escalation Cohort 2a | Phase 1b Dose Escalation Cohorts 1, 2b and 2c | Phase 1b Dose Escalation Cohort 3 | Phase 2 RP2D - Capsule | Phase 2 RP2D - Tablet
Number analyzed (Participants) | 5 | 15 | 5 | 30 | 9
ng/mL
  Single-dose: number analyzed (Participants) | 5 | 15 | 4 | 27 | 8
  Single-dose | 29.8 (26.7) | 83.3 (38.1) | 214 (140) | 196 (166) | 298 (137)
  Multiple-dose: number analyzed (Participants) | 0 | 0 | 0 | 9 | 8
  Multiple-dose |  |  |  | 334 (283) | 238 (208)

10. Secondary Outcome: Cmax (ng/mL) of Valganciclovir
Description: PK assessment of valganciclovir pre-dose and at hours 0.5, 1, 2, 4, and 6 post-dose on C1D1 and C2D1
Time Frame: Phase 1b: Cycle 1 Day 1 and Phase 2: multiple doses through Cycle 2 Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Phase 1b Dose Escalation - 450 mg: valganciclovir: 450 mg QD or BID VRx-3996: 5 mg BID, 10 mg QD or BID
- Phase 1b Dose Escalation - 900 mg: valganciclovir: 900mg QD or BID VRx-3996: 10 mg QD or BID, 20 mg QD on Days 1 to 4/week
- Phase 2 RP2D - Capsule (VRx-3996); Phase 2 RP2D - Tablet (VRx-3996): valganciclovir: 900 mg QD VRx-3996: 20 mg QD on Days 1 to 4/week
Arm/Group | Phase 1b Dose Escalation - 450 mg | Phase 1b Dose Escalation - 900 mg | Phase 2 RP2D - Capsule (VRx-3996) | Phase 2 RP2D - Tablet (VRx-3996)
Number analyzed (Participants) | 13 | 12 | 30 | 9
ng/mL
  Single-Dose | 4230 (1348) | 6712 (1495) | 7300 (2790) | 14900 (8380)
  Multiple-Dose: number analyzed (Participants) | 0 | 0 | 11 | 8
  Multiple-Dose |  |  | 8690 (5800) | 14200 (7060)

11. Secondary Outcome: Area Under Curve (AUC) 0-t of VRx-3996
Description: PK assessment of VRx-3996 pre-dose and at hours 0.5, 1, 2, 4, and 6 post-dose on C1D1 and C2D1
Time Frame: Phase 1b: Cycle 1 Day 1 and Phase 2: multiple doses through Cycle 2 Day 1
Population: The PK Analysis Set was used for all PK analyses and included all patients in the intent-to-treat population (defined as all enrolled patients) who had at least one postdose measurable PK concentration. The PK Analysis Set will be used for individual plasma concentration listings and summaries of plasma concentrations. The PK Population will also be used for individual and mean figures for plasma concentrations.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Phase 1b Dose Escalation Cohort 2a | Phase 1b Dose Escalation Cohorts 1, 2b and 2c | Phase 1b Dose Escalation Cohort 3 | Phase 2 RP2D - Capsule | Phase 2 RP2D - Tablet
Number analyzed (Participants) | 5 | 15 | 5 | 30 | 9
h*ng/mL
  Single-dose: number analyzed (Participants) | 3 | 14 | 2 | 26 | 7
  Single-dose | 128 (67.0) | 229 (76.4) | 340 (384) | 417 (299) | 587 (212)
  Multiple-dose: number analyzed (Participants) | 0 | 0 | 0 | 8 | 7
  Multiple-dose |  |  |  | 638 (418) | 474 (268)

12. Secondary Outcome: AUC 0-t of of Valganciclovir
Description: PK assessment of valganciclovir pre-dose and at hours 0.5, 1, 2, 4, and 6 post-dose on C1D1 and C2D1
Time Frame: Phase 1b: Cycle 1 Day 1 and Phase 2: multiple doses through Cycle 2 Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Phase 1b Dose Escalation - 450 mg | Phase 1b Dose Escalation - 900 mg | Phase 2 RP2D - Capsule (VRx-3996) | Phase 2 RP2D - Tablet (VRx-3996)
Number analyzed (Participants) | 13 | 12 | 30 | 9
h*ng/mL
  Single-dose: number analyzed (Participants) | 12 | 11 | 29 | 7
  Single-dose | 15600 (4160) | 24400 (9300) | 25200 (10400) | 49700 (29100)
  Multiple-dose: number analyzed (Participants) | 0 | 0 | 11 | 8
  Multiple-dose |  |  | 28300 (16400) | 46600 (18000)

13. Secondary Outcome: Half-life of VRx-3996
Description: PK assessment of VRx-3996 pre-dose and at hours 0.5, 1, 2, 4, and 6 post-dose on C1D1 and C2D1
Time Frame: Phase 1b: Cycle 1 Day 1 and Phase 2: multiple doses through Cycle 2 Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 1b Dose Escalation Cohort 2a | Phase 1b Dose Escalation Cohorts 1, 2b and 2c | Phase 1b Dose Escalation Cohort 3 | Phase 2 RP2D - Capsule | Phase 2 RP2D - Tablet
Number analyzed (Participants) | 5 | 15 | 5 | 30 | 9
hours
  Single-dose: number analyzed (Participants) | 5 | 13 | 0 | 16 | 8
  Single-dose | 1.89 (0.252) | 1.44 (0.466) |  | 1.46 (0.589) | 1.43 (0.287)
  Multiple-dose: number analyzed (Participants) | 0 | 0 | 0 | 5 | 6
  Multiple-dose |  |  |  | 1.10 (0.181) | 1.87 (1.33)

14. Secondary Outcome: Half-life of Valganciclovir
Description: PK assessment of valganciclovir pre-dose and at hours 0.5, 1, 2, 4, and 6 post-dose on C1D1 and C2D1
Time Frame: Phase 1b: Cycle 1 Day 1 and Phase 2: multiple doses through Cycle 2 Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 1b Dose Escalation - 450 mg | Phase 1b Dose Escalation - 900 mg | Phase 2 RP2D - Capsule (VRx-3996) | Phase 2 RP2D - Tablet (VRx-3996)
Number analyzed (Participants) | 11 | 10 | 23 | 6
hours
  Single-dose | 3.56 (1.06) | 3.13 (1.43) | 3.32 (1.10) | 2.17 (1.68)
  Multiple-dose: number analyzed (Participants) | 0 | 0 | 7 | 5
  Multiple-dose |  |  | 2.43 (0.697) | 2.61 (1.55)

ADVERSE EVENTS:
Time Frame: Up to approximately 2 years
Description: Valganciclovir dosage reductions were allowed for participants with renal impairment at study entry or during study treatment.
Arm/Group | Phase 1b Dose Escalation Cohort 1 | Phase 1b Dose Escalation Cohort 2a | Phase 1b Dose Escalation Cohort 2b | Phase 1b Dose Escalation Cohort 2c | Phase 1b Dose Escalation Cohort 3 | Phase 2 Dose Expansion - Capsule | Phase 2 Dose Expansion - Tablet
All-Cause Mortality (participants affected / at risk) | 4/7 | 4/5 | 2/4 | 4/4 | 3/5 | 17/30 | 4/9
Serious Adverse Events (participants affected / at risk) | 2/7 | 2/5 | 2/4 | 1/4 | 1/5 | 11/30 | 4/9
Other Adverse Events (participants affected / at risk) | 7/7 | 5/5 | 4/4 | 4/4 | 5/5 | 22/30 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b Dose Escalation Cohort 1 (N=7) | Phase 1b Dose Escalation Cohort 2a (N=5) | Phase 1b Dose Escalation Cohort 2b (N=4) | Phase 1b Dose Escalation Cohort 2c (N=4) | Phase 1b Dose Escalation Cohort 3 (N=5) | Phase 2 Dose Expansion - Capsule (N=30) | Phase 2 Dose Expansion - Tablet (N=9)
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterocolitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b Dose Escalation Cohort 1 (N=7) | Phase 1b Dose Escalation Cohort 2a (N=5) | Phase 1b Dose Escalation Cohort 2b (N=4) | Phase 1b Dose Escalation Cohort 2c (N=4) | Phase 1b Dose Escalation Cohort 3 (N=5) | Phase 2 Dose Expansion - Capsule (N=30) | Phase 2 Dose Expansion - Tablet (N=9)
Thrombocytopenia (Gastrointestinal disorders) | 2 | 2 | 0 | 2 | 0 | 5 | 0
Constipation (Gastrointestinal disorders) | 1 | 4 | 0 | 2 | 2 | 8 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 2 | 0 | 1 | 7 | 4
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 2 | 6 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 3 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 4 | 1 | 0 | 0 | 1 | 10 | 6
Pyrexia (General disorders) | 0 | 2 | 2 | 0 | 1 | 6 | 2
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Oedema peripheral (General disorders) | 4 | 0 | 0 | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 2 | 0 | 0 | 0 | 5 | 3
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 1 | 1 | 2 | 11 | 4
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 5 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 6 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 4 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 3 | 0 | 0 | 3 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 1 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 3 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 0 | 1 | 5 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 3 | 1 | 4 | 11 | 5
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 3 | 1 | 0 | 0 | 3 | 3 | 1
Platelet count decreased (Investigations) | 3 | 0 | 1 | 0 | 0 | 3 | 3
White blood cell count decreased (Investigations) | 2 | 1 | 1 | 0 | 0 | 4 | 3
Lymphocyte count decreased (Investigations) | 2 | 1 | 0 | 0 | 0 | 3 | 2
Weight decreased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyoderma (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 6 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT03397706/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT03397706/SAP_001.pdf